CLINICAL TRIAL: NCT00006223
Title: A Phase III Study of Flt3 Ligand (Flt3L) Therapy in Acute Myeloid Leukemia (AML) Patients in Remission
Brief Title: flt3L in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); SWOG Cancer Research Network (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068143; ECOG-2998; CALGB-19903; SWOG-E2998
Record Dates: First submitted 2000-09-11; First posted 2003-09-03 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2006-09

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute promyelocytic leukemia (M3); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); adult acute monocytic leukemia (M5b); adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — flt3 ligand protein

INTERVENTIONS:
Biological: recombinant flt3 ligand

SUMMARY:
RATIONALE: Drugs such as flt3L may stimulate a person's immune system and help kill cancer cells. It is not yet known if flt3L is effective in treating acute myeloid leukemia.

PURPOSE: Randomized phase III trial to determine the effectiveness of flt3L in treating patients who have acute myeloid leukemia that is in remission.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the failure-free survival and overall survival in patients with acute myeloid leukemia in complete remission treated with maintenance flt3 ligand vs observation alone.
* Compare the long-term immunologic effects of these regimens in these patients.
* Compare the long-term safety and toxicity of these regimens in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to complete remission (CR) (first vs second vs third or subsequent) and post-remission therapy (yes vs no). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive flt3 ligand subcutaneously daily on days 1-14. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo observation alone. Patients begin treatment or observation within 4 weeks after documentation of CR after induction therapy or within 4 weeks after discharge from hospital after post-remission therapy.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 139 patients will be accrued for this study within approximately 28 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia in first, second, third, or subsequent complete remission (CR)

  * Must be at least 60 years of age if first CR
  * Must have had histological proof (from bone marrow aspirate, smears, or touch preps of marrow biopsy) of one of the following prior to achieving CR:

    * Acute myeloblastic leukemia (M0, M1, M2)
    * Acute promyelocytic leukemia (M3)
    * Acute myelomonocytic leukemia (M4)
    * Acute monocytic leukemia (M5)
    * Acute erythroleukemia (M6)
    * Acute megakaryocytic leukemia (M7)
    * Refractory anemia with excess blasts in transformation

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 3 times upper limit of normal (ULN)
* SGOT less than 3 times ULN

Renal:

* Creatinine less than 2 mg/dL

Cardiovascular:

* No clinically significant active cardiac disease

Pulmonary:

* No clinically significant active pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No uncontrolled or active autoimmune disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior autologous bone marrow transplantation (BMT) allowed
* No prior allogeneic BMT
* Other prior immunotherapy allowed if not received during the most recent treatment

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob M. Rowe, MD, Study Chair — Rambam Health Care Campus; Richard A. Larson, MD, Study Chair — University of Chicago; John E. Godwin, MD, MS, Study Chair — Loyola University
Locations (47):
- United States (47):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia